CLINICAL TRIAL: NCT02139384
Title: Development of a Clinical Pediatric Pneumonia Score in Critically Ill Children Admitted With Acute Respiratory Failure
Brief Title: Clinical Pediatric Pneumonia Score in Critically Ill Children
Status: Withdrawn | Type: Observational
Why Stopped: The study was withdrawn due to inability to enroll patients in a timely fashion.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5110327
Record Dates: First submitted 2014-05-08; First posted 2014-05-15 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Community Acquired Pneumonia
Keywords: procalcitonin; community acquired pneumonia; pneumonia score
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to create a clinical pneumonia tool that can be used to predict the cause of community-acquired pneumonia, which is a lung infection that began outside of the hospital in critically ill children therefore limiting unnecessary antibiotic use. The investigators will enroll critically ill children admitted with acute respiratory failure and suspected pneumonia. Each patient will receive a clinical pneumonia score blinded from culture and respiratory viral panel results. All care after samples obtained will be at the discretion of the PICU team. The investigators believe that our clinical pneumonia scale with procalcitonin will accurately designate viral from bacterial etiologies.

ELIGIBILITY:
Inclusion Criteria:

* All intubated pediatric patients
* Age 1 day to 21 years
* Admitted to the LLUCH PICU with suspected pneumonia for the next 6 months
* Have received antibiotics for less than 12 hours
* Have been intubated for less than 24 hours
* Patients must be English or Spanish speaking for consent purposes.

Exclusion Criteria:

* Patients who have received antibiotics for greater than 12 hours
* Patients who have been intubated for greater than 24 hours
* Patients who are unable to tolerate non-bronchoscopic bronchoalveolar lavage

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: critically ill children admitted the the LLU PICU with acute respiratory failure with suspected community-acquired pneumonia
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Can our proposed pneumonia score distinguish community acquired bacterial pneumonia from community acquired viral pneumonia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Tinsley, M.D., Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Children's Hospital, Loma Linda, California, United States